CLINICAL TRIAL: NCT02522143
Title: College Students Who Self-Harm: An Intervention Study
Brief Title: College Students Who Self-Harm
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1310M45125
Record Dates: First submitted 2014-02-07; First posted 2015-08-13 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Borderline Personality Disorder; Suicide
Keywords: self-harm; self-mutilation; cutting
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Informational Sessions (Sham Comparator): Control intervention consists of informational sessions describing BPD characteristics/ treatment and time- / stress-management skills
  Interventions: Behavioral: Informational sessions describing BPD characteristics
- Condensed-DBT treatment intervention (Experimental): Condensed-DBT treatment intervention includes all DBT components, tailored to students.
  Interventions: Behavioral: Condensed-DBT treatment intervention

INTERVENTIONS:
Behavioral: Informational sessions describing BPD characteristics — Control intervention consists of informational sessions describing BPD characteristics/ treatment and time- / stress-management skills
  Arms: Informational Sessions
Behavioral: Condensed-DBT treatment intervention — The Intervention consists of an 8-week manual based psychoeducational group utilizing modified condensed-DBT Treatment manual previously used in a treatment study (Moen et al, 2012).
  Other Names: The proposed Condensed-DBT treatment intervention includes all DBT components, tailored to students.
  Arms: Condensed-DBT treatment intervention

SUMMARY:
Study Aims/Objectives:

This projects' Primary Aim is development of a Condensed DBT Stepped Care Model tailored to the unique requirements of students meeting sub-clinical diagnostic criteria for BPD (Borderline Personality Disorder) with its associated high rate of self-harm and suicide.

DETAILED DESCRIPTION:
Study Aims/Objectives:

This projects' Primary Aim is development of a Condensed DBT Stepped Care Model tailored to the unique requirements of students meeting sub-clinical diagnostic criteria for BPD with its associated high rate of self-harm and suicide. The investigator previously implemented a 4-mth condensed-DBT regimen with success in an adult clinical population. This study will evaluate an intensive 8 week intervention formulated for students to reduce the high prevalence of self-harm and dysfunctional behavior in this population and reduce the need for extended treatment in later years. It will include rigorous screening for collateral disorders, including Substance Use Disorders exacerbating BPD symptoms and suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 27
* Currently enrolled in college
* Meet at least 4 of 9 Criteria of BPD (DSM-V) with one criterion being self-harm (e.g. cut, burn, or hit self)

Exclusion Criteria:

* have a current major psychiatric disorder diagnosis, or other gross cognitive impairment (as identified in the phone screen or the SCID I measure) or
* have undergone DBT or
* are suicidal and require full DBT and/or hospitalization or
* are currently in any other individual or group therapy
* unable to attend weekly visits over 8 weeks, starting March 24, 2014

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in BPD (Borderline Personality Disorder) behaviors | 8-weeks
  produce greater decreases in depression, anxiety, self-harm, and other BPD behaviors,

SECONDARY OUTCOMES:
Change in reported psychiatric symptoms, | 8-weeks
  diminish reported psychiatric symptoms, and Decreased utilization of Emergency Room, crisis, and University Disability Services on campus.
Diminished emergency room visits | 8 weeks
  self reported ER visits

CONTACTS AND LOCATIONS:
Overall Officials: Richelle N Moen,, PhD, Principal Investigator — University of Minnesota
Locations (1):
- CTSI, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617